CLINICAL TRIAL: NCT03089372
Title: Low Intensity Extracorporeal Shock Wave Treatment (LI-ESWT) in Patients With Vasculogenic Erectile Dysfunction (ED): Evaluation of the Efficacy of Re-treatment.
Brief Title: Effect of Repeating Low Intensity Extracorporeal Shock Wave Treatment (LI-ESWT) for Erectile Dysfunction (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases, Greece
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4240/2016
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Low intensity extracorporeal shock wave treatment
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive two sessions of LI-ESWT per week for a 3 week period (6 sessions totally)
  Interventions: Device: ARIES-ED device
- Group B (Active Comparator): Patients will receive one session of LI-ESWT per week for a 6 week period (6 sessions totally)
  Interventions: Device: ARIES-ED device

INTERVENTIONS:
Device: ARIES-ED device — The Dornier Aries-ED device will be used for the purpose of the study. LI-ESWT will be applied to the penile shaft 3 areas, and the 2 crura (two sites).

SUMMARY:
The present study evaluates the efficacy and safety of repetitive treatments of Low Intensity Extracorporeal Shock Wave Treatment (LI-ESWT) using Aries ED device in men with mild-moderate and severe vasculogenic ED, who have previously responded to oral PDE5-Is, and completed 6 or 12 sessions of LI-ESWT with Aries device during the last 6 month.

DETAILED DESCRIPTION:
This is an extension, 2 parallel arms, clinical trial of a previous study in which patients were PDE5I users/responders and were randomized to receive either one or two shockwave treatment sessions per week for a total of 6 weeks, without treatment interval. After completing the 6-month follow up of the first trial , ED patients will be screened, in order to identify if the IIEF ED domain is still abnormal (<26). Afterwards, the 2 groups of the first study will follow the 2 different treatment protocols (once vs twice per week). All patients will receive 6 treatment sessions with Aries, with the same energy level. First treatment session will take place between days 0-28 from the day of the 6-month follow up. All patients will agree and sign a new Informed Consent Form. Therefore, patients who took 6 sessions once a week (Group A in the previous trial) will be switched to take 6 sessions twice a week in 3 weeks, and those already treated with 12 sessions twice a week (Group B in the previous trial) will be treated with 6 sessions once a week.

Study visits and duration

Baseline - Visit: the basic work-up will take place, including medical and sexual history, as well as lab tests, if indicated by medical history. The IIEF-ED domain will be measured, as well as the Sexual Encounter Profile (SEP) for the last 4-week period with at least 4 attempts for intercourse (without PDE5i use). The study criteria will be checked and if patients are eligible (IIEF-ED domain <26), they will receive their first repetitive treatment, either on the same day as the 6-month follow up of the previous study or within maximum 4 weeks.

Treatment Visits: In all treatment visits, patients will receive active LI-ESWT treatment, according to the study protocol. Group A will receive treatment twice per week for three weeks and Group B will receive treatment once per week for six weeks. Interval between 2 treatments will be 7+2days for Group B and 3+1 day for Group A. Adverse events and changes in concomitant medication will be recorded. PDE5i intake is prohibited throughout the treatment period.At visit 6 penile ultrasonography will be conducted in order to check for potential adverse events related to the treatment.

Follow-up visit 1 - 3 (4, 12 and 24 weeks post treatment): the SEP diaries will be returned and the IIEF-ED domain will be completed for the 4 weeks prior to the aforementioned timepoints, during which no PDE5i intake is allowed. The document of the visit (protocol compliance, adverse events) will be completed. At week 12, triplex ultrasonography will be performed by the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate
2. Age >18
3. Presence of vasculogenic erectile dysfunction for at least 6 months
4. Positive response to PDE5i
5. Patients who completed the 6 months follow-up of a previous study including 6 or 12 sessions of LI-ESWT with Aries device and still have an abnormal IIEF ED domain (< 26)
6. Abnormal penile triplex-based hemodynamic parameters (peak flow velocity <35cm/sec)
7. Stable heterosexual relationship for more than 3 months
8. Sexually active and agree to suspend all ED therapy for the duration of study

Exclusion Criteria:

1. Any cause of ED other than vascular related
2. Previous radiation therapy to pelvis
3. History of radical prostatectomy
4. Clinically significant chronic haematological disease
5. Cardiovascular conditions that prevent sexual activity
6. Peyronie's Disease or penile curvature
7. History of heart attack, stroke or any life- threatening arrhythmia within the prior 6 month
8. Anti-androgens oral or injectables androgens
9. Untreated Hypogonadism as demonstrated by abnormal testosterone levels
10. Malignancy within the past 5 years
11. Any unstable medical, psychiatric condition or spinal cord injury
12. Anatomical or neurological abnormalities in the treatment area
13. Use of any treatment for ED within 7 days of screening ( oral medications, vacuum devices, constrictive devices, injections or urethral suppositories)
14. Known allergy to ultrasound gel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
The percent of subjects who achieve clinically important difference (MCID) in the EF domain score of the IIEF | at 6 month follow up visit.
  MCID is defined according to baseline ED severity as:
  * Improvement by 2 or more in the EF domain score of the IIEF for patients with mild ED ( EF scores 17-25) at baseline.
  * Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED(EF scores 11-16) at baseline
  * Improvement by 7 or more in the EF domain score of the IIEF for patients with severe ED (EF scores 0-10) at baseline

SECONDARY OUTCOMES:
Change in the EF domain score of the IIEF | baseline and 6 month follow up visit
  EF domain of the IIEF questionnaire will be completed
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 6 month follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
Change in mean peak systolic velocity (PSV) | baseline and 3 month follow up visit
  Mean peak systolic velocity will be measured by penile triplex ultrasonography by the same investigator.
Number of patients with treatment related adverse events | 27 months (Group A) ,30 months (Group B)
  Potential treatment related adverse events after the first LI-ESWT session and during the 6 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases (ISUD)
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Z, Lin G, Reed-Maldonado A, Wang C, Lee YC, Lue TF. Low-intensity Extracorporeal Shock Wave Treatment Improves Erectile Function: A Systematic Review and Meta-analysis. Eur Urol. 2017 Feb;71(2):223-233. doi: 10.1016/j.eururo.2016.05.050. Epub 2016 Jun 16. PMID 27321373
- [Background] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Gruenwald I, Kitrey ND, Appel B, Vardi Y. Low-Intensity Extracorporeal Shock Wave Therapy in Vascular Disease and Erectile Dysfunction: Theory and Outcomes. Sex Med Rev. 2013 Jul;1(2):83-90. doi: 10.1002/smrj.9. Epub 2015 Oct 18. PMID 27784587
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209